CLINICAL TRIAL: NCT01476787
Title: A Phase 3 Open-Label Randomized Study to Compare the Efficacy and Safety of Rituximab Plus Lenalidomide (CC-5013) Versus Rituximab Plus Chemotherapy in Subjects With Previously Untreated Follicular Lymphoma
Brief Title: Combined Rituximab and Lenalidomide Treatment for Untreated Patients With Follicular Lymphoma
Acronym: RELEVANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-FOL-GELARC-0683C; 2011-002792-42 (EudraCT Number)
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Follicular Lymphoma
Keywords: Follicular lymphoma; Non-Hodgkins Follicular Lymphoma; treatment for Follicular Lymphoma; rituximab treatment; rituximab and lenalidomide treatment
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide + Rituximab (Experimental): * Lenalidomide dose 20-mg on days 2-22 every 28 days for 6 cycles, if CR then 10-mg on days 2-22 every 28 days for 12 cycles. PR after 6 cycles, continue 20 mg for 3~6 cycles and then 10 mg on days 2-22 every 28-day cycles for up to 18 cycles.
  * Rituximab, 375 mg/m2 on days 1, 8, 15 and 22 of cycle 1, day 1 of cycles 2 to 6; 8 weeks later responding patients continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Interventions: Drug: Rituximab; Drug: Lenalidomide
- Control (Active Comparator): • ONE of the following: Rituximab-CHOP, Rituximab-CVP, Rituximab-Bendamustine. 7 to 8 weeks later responding patients will continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Interventions: Drug: Rituximab-CHOP; Drug: Rituximab-CVP; Drug: Rituximab-Bendamustine

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 on days 1, 8, 15 and 22 of cycle 1, day 1 of cycles 2 to 6; 8 weeks later responding patients continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Arms: Lenalidomide + Rituximab
Drug: Lenalidomide — 20-mg on days 2-22 every 28 days x 6 cycles, if CR then 10-mg on days 2-22 every 28 days for 12 cycles. PR after 6 cycles, continue 20 mg for 3~6 cycles and then 10 mg on days 2-22 every 28-day cycles for upto 18 cycles
  Other Names: Revlimid
  Arms: Lenalidomide + Rituximab
Drug: Rituximab-CHOP — 7 to 8 weeks later responding patients will continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Arms: Control
Drug: Rituximab-CVP — 7 to 8 weeks later responding patients will continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Arms: Control
Drug: Rituximab-Bendamustine — 7 to 8 weeks later responding patients will continue with 375 mg/m2 rituximab every 8 weeks for 12 cycles.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effect of the combined treatment of lenalidomide and rituximab in controlling the Follicular Lymphoma disease and also increase the length of response compared to the available standard combination chemotherapy treatment for Follicular Lymphoma.

DETAILED DESCRIPTION:
Follicular Lymphoma (FL) is a cancer of a B lymphocyte, a type of white blood cell. FL is typically a slowly progressing but incurable disease. Follicular lymphoma cells produce a specific defect in the patient's immune system impairing their ability to control their cancer. Lenalidomide has been shown to reverse the specific immune defect caused by FL in the patient. By including lenalidomide, the RELEVANCE study aims to eliminate the cancer while restoring the patient's immune competence.

The 'Relevance' cooperative group trial is being conducted as two companion studies: RV-FOL-GELARC-0683 (N=750) and RV-FOL-GELARC-0683C (N=250); the combined total of 1000 Follicular Lymphoma patients enrolled in both studies will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma grade 1, 2 or 3a, Stage II-IV
* Have no prior systemic treatment for lymphoma
* Symptomatic follicular lymphoma requiring treatment.
* Age ≥18 years
* Eastern Cooperative oncology group performance status 0-2
* Willing to follow pregnancy precautions

Exclusion Criteria:

* Clinical evidence of transformed lymphoma or Grade 3b follicular lymphoma.
* Major surgery (excluding lymph node biopsy) within 28 days prior to signing informed consent.
* Known seropositive for or active viral infection with hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV)
* Known sensitivity or allergy to murine products.
* Presence or history of central nervous system involvement by lymphoma
* At high risk for a venous thromboembolic event (VTE) and not willing to take VTE prophylaxis
* Any of the following laboratory abnormalities:
* serum aspartate transaminase or alanine transaminase > 3x upper limit of normal (ULN), except in patients with documented liver involvement by lymphoma
* total bilirubin > 2.0 mg/dl (34 µmol/L) except in cases of Gilberts Syndrome and documented liver or pancreatic involvement by lymphoma
* creatinine clearance of < 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2011-12-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Morschhauser, MD, PhD, Study Chair — The Lymphoma Study Association (LYSA)
Locations (36):
- United States (26):
  - Local Institution - 54103, Chandler, Arizona
  - Local Institution - 51803, Fullerton, California
  - Local Institution - 52003, Los Angeles, California
  - Local Institution - 51603, Colorado Springs, Colorado
  - Local Institution - 52503, Englewood, Florida
  - Local Institution - 51703, Orlando, Florida
  - Local Institution - 53803, St. Petersburg, Florida
  - Local Institution - 50803, Chicago, Illinois
  - Local Institution - 52203, Lexington, Kentucky
  - Local Institution - 53603, Westminster, Maryland
  - Local Institution - 50403, Boston, Massachusetts
  - Local Institution - 50503, Boston, Massachusetts
  - Local Institution - 53003, Southfield, Michigan
  - Local Institution - 51003, St Louis, Missouri
  - Local Institution - 54403, Cherry Hill, New Jersey
  - Local Institution - 53703, Hackensack, New Jersey
  - Local Institution - 50903, Morristown, New Jersey
  - Local Institution - 54303, Sparta, New Jersey
  - Local Institution - 52403, New York, New York
  - Local Institution - 50203, New York, New York
  - Local Institution - 51303, Nashville, Tennessee
  - Local Institution - 51203, Dallas, Texas
  - Local Institution - 51103, Houston, Texas
  - Local Institution - 54003, Lubbock, Texas
  - Local Institution - 53303, Richmond, Virginia
  - Local Institution - 52703, Seattle, Washington
- Japan (10):
  - Local Institution - 40722, Chuo-ku, Tokyo
  - Local Institution - 40222, Koto-ku, Tokyo
  - Local Institution - 41122, Minato-ku, Tokyo
  - Local Institution - 40922, Fukuoka
  - Local Institution - 40422, Hiroshima
  - Local Institution - 40122, Isehara City, Kanagawa
  - Local Institution - 40322, Kobe
  - Local Institution - 40622, Kyoto
  - Local Institution - 41022, Sendai
  - Local Institution - 40522, Shizuoka

REFERENCES:
- [Background] Morschhauser F, Fowler NH, Feugier P, Bouabdallah R, Tilly H, Palomba ML, Fruchart C, Libby EN, Casasnovas RO, Flinn IW, Haioun C, Maisonneuve H, Ysebaert L, Bartlett NL, Bouabdallah K, Brice P, Ribrag V, Daguindau N, Le Gouill S, Pica GM, Martin Garcia-Sancho A, Lopez-Guillermo A, Larouche JF, Ando K, Gomes da Silva M, Andre M, Zachee P, Sehn LH, Tobinai K, Cartron G, Liu D, Wang J, Xerri L, Salles GA; RELEVANCE Trial Investigators. Rituximab plus Lenalidomide in Advanced Untreated Follicular Lymphoma. N Engl J Med. 2018 Sep 6;379(10):934-947. doi: 10.1056/NEJMoa1805104. PMID 30184451
- [Background] Fowler NH, Davis RE, Rawal S, Nastoupil L, Hagemeister FB, McLaughlin P, Kwak LW, Romaguera JE, Fanale MA, Fayad LE, Westin JR, Shah J, Orlowski RZ, Wang M, Turturro F, Oki Y, Claret LC, Feng L, Baladandayuthapani V, Muzzafar T, Tsai KY, Samaniego F, Neelapu SS. Safety and activity of lenalidomide and rituximab in untreated indolent lymphoma: an open-label, phase 2 trial. Lancet Oncol. 2014 Nov;15(12):1311-8. doi: 10.1016/S1470-2045(14)70455-3. Epub 2014 Oct 15. PMID 25439689
- [Background] Ahmadi T, Chong EA, Gordon A, Aqui NA, Nasta SD, Svoboda J, Mato AR, Schuster SJ. Combined lenalidomide, low-dose dexamethasone, and rituximab achieves durable responses in rituximab-resistant indolent and mantle cell lymphomas. Cancer. 2014 Jan 15;120(2):222-8. doi: 10.1002/cncr.28405. Epub 2013 Oct 7. PMID 24122387
- [Background] Delfau-Larue MH, Boulland ML, Beldi-Ferchiou A, Feugier P, Maisonneuve H, Casasnovas RO, Lemonnier F, Pica GM, Houot R, Ysebaert L, Tilly H, Eisenmann JC, Le Gouill S, Ribrag V, Godmer P, Glaisner S, Cartron G, Xerri L, Salles GA, Fest T, Morschhauser F. Lenalidomide/rituximab induces high molecular response in untreated follicular lymphoma: LYSA ancillary RELEVANCE study. Blood Adv. 2020 Aug 11;4(14):3217-3223. doi: 10.1182/bloodadvances.2020001955. PMID 32673385
- [Derived] Laurent C, Trisal P, Tesson B, Seth S, Beyou A, Roulland S, Lesne B, Van Acker N, Cerapio JP, Chartier L, Guille A, Stokes ME, Huang CC, Huet S, Gandhi AK, Morschhauser F, Xerri L. Follicular lymphoma comprises germinal center-like and memory-like molecular subtypes with prognostic significance. Blood. 2024 Dec 12;144(24):2503-2516. doi: 10.1182/blood.2024024496. PMID 39374535
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1030 participants were randomized, 1010 participants were treated.
Groups:
- Rituximab-Lenalidomide: Rituximab, 375 mg/m^2 on days
  1, 8, 15 and 22 of cycle 1, day 1 of cycles 2 to 6; and 8 weeks later responding patients continue with 375 mg/m^2 rituximab every 8 weeks for 12 cycles. Six cycles of lenalidomide 20 mg daily on days 2-22 every 28 days.
- Investigator Choice: Rituximab-CHOP: with six cycles of R-CHOP in 21 day cycles followed by two 21 day cycles of 375 mg/m^2 rituximab and 7 weeks later responding patients continue with 375 mg/m^2 rituximab every 8 weeks for 12 cycles, OR Rituximab-CVP: with eight cycles of R-CVP in 21 day cycles; and 7 weeks later responding patients continue with 375 mg/m^2 rituximab every 8 weeks for 12 cycles, OR Rituximab-Bendamustine: with rituximab 375 mg/m^2 (day 1) plus bendamustine 90 mg/m^2 (days 1 + 2) every 28 days for six cycles; and 8 weeks later responding patients continue with 375 mg/m^2 rituximab every 8 weeks for 12 cycles.
Period: Pre-treatment
Arm/Group | Rituximab-Lenalidomide | Investigator Choice
Started | 513 | 517
Completed | 507 | 503
Not Completed | 6 | 14
Period: Treatment
Arm/Group | Rituximab-Lenalidomide | Investigator Choice
Started | 507 | 503
Completed | 350 | 357
Not Completed | 157 | 146
Not completed — Progression | 64 | 71
Not completed — Toxicity | 44 | 16
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 3 | 14
Not completed — Major protocol violation | 1 | 6
Not completed — Other reasons | 10 | 22
Not completed — Concurrent illness | 12 | 9
Not completed — Insufficient response | 15 | 3
Not completed — Voluntary treatment discontinuation | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab-Lenalidomide | Investigator Choice | Total
Number analyzed (Participants) | 513 | 517 | 1030
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (11.23) | 58.3 (11.38) | 58.4 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262 | 266 | 528
  Male | 251 | 251 | 502
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CR/CRu) at 120 Weeks by Independent Central Review
Description: The Complete Response Rate (CR/CRu) is the percentage of participants who achieve complete response (CR/CRu) at 120 weeks as assessed per Independent Central Review.
  * Complete Response (CR): Disappearance of all evidence of disease.
  * Complete Response Unconfirmed (CRu): Disappearance of all disease with the exception of residual lymph nodes that are 1.5 cm or less in greatest transverse diameter and/or indeterminate bone marrow findings.
Time Frame: At 120 weeks
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Rituximab-Lenalidomide | Investigator Choice
Number analyzed (Participants) | 513 | 517
Percent of participants | 48.1 [43.7 to 52.6] | 53.0 [48.6 to 57.4]
Statistical Analysis 1: Comparison: Rituximab-Lenalidomide vs Investigator Choice; Test type: Superiority; p = 0.128, Cochran-Mantel-Haenszel

2. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from randomization into the study to the first observation of documented disease progression or death due to any cause.
  Progressive Disease (PD) is characterized by any of the following:
  * An increase of at least 50% in the sum of the products of the greatest diameters (SPD) of any previously identified abnormal lymph node(s) or other disease sites.
  * The appearance of any new lesion during or after treatment.
  * An increase of at least 50% in the longest diameter of a previously identified node that was 1 cm or more in its short axis.
  * An increase of at least 50% in the size of other lesions (e.g., splenomegaly, hepatomegaly).
  Based on Kaplan-Meier estimates.
Time Frame: From randomization into the study to the first observation of documented disease progression or death due to any cause (up to approximately 140 months).
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab-Lenalidomide | Investigator Choice
Number analyzed (Participants) | 513 | 517
Months | 120.2 [104.9 to 126.3] | 123.8 [107.4 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Rituximab-Lenalidomide vs Investigator Choice; Test type: Superiority; p = 0.406, Log Rank; Hazard Ratio (HR) = 0.920, 95% CI 2-sided [0.756 to 1.120]

3. Secondary Outcome: Complete Response Rate (CR) at 120 Weeks Per Independent Central Review
Description: The Complete Response Rate (CR) is the percentage of participants who achieve confirmed complete response (CR) at 120 weeks as assessed per Independent Central Review.
  - Complete Response (CR): Disappearance of all evidence of disease.
Time Frame: At 120 weeks
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Rituximab-Lenalidomide | Investigator Choice
Number analyzed (Participants) | 513 | 517
Percent of participants | 27.7 [23.8 to 31.8] | 32.7 [28.7 to 36.9]

4. Secondary Outcome: Event-free Survival (EFS)
Description: Event Free Survival (EFS) is defined as the time a participant remains free from certain negative events (disease progression, relapse, initiation of a new anti-lymphoma treatment, or death) between the date of randomization to the date of first documented progression, relapse, and initiation of a new anti-lymphoma treatment or death by any cause. Responding participants and those lost to follow up were censored at their last tumor assessment date.
  Progressive Disease (PD) is characterized by any of the following:
  * An increase of at least 50% in the sum of the products of the greatest diameters (SPD) of any previously identified abnormal lymph node(s) or other disease sites.
  * The appearance of any new lesion during or after treatment.
  * An increase of at least 50% in the longest diameter of a previously identified node that was 1 cm or more in its short axis.
  * An increase of at least 50% in the size of other lesions (e.g., splenomegaly, hepatomegaly).
  Based on Kaplan-Meier estimates.
Time Frame: From randomization to the date of first documented progression, relapse, and initiation of a new anti-lymphoma treatment or death by any cause (up to approximately 140 months).
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab-Lenalidomide | Investigator Choice
Number analyzed (Participants) | 513 | 517
Months | 130.6 [121.9 to NA] — Insufficient number of participants with events | 132.3 [115.7 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Rituximab-Lenalidomide vs Investigator Choice; Test type: Superiority; Hazard Ratio (HR) = 1.038, 95% CI 2-sided [0.854 to 1.261]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the median length of time a participant stays alive from randomization. Participants who died, regardless of the cause of death, were considered to have had an event. Participants who withdrew consent for the study were considered censored at the time of withdrawal. Participants who completed the study and were still alive at the time of the clinical data cut-off date were censored. All participants who were lost to follow-up prior to the clinical data cut-off date were also considered censored at the time of last contact. Based on Kaplan-Meier estimates.
Time Frame: From randomization to the date of death by any cause (up to approximately 144 months).
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab-Lenalidomide | Investigator Choice
Number analyzed (Participants) | 513 | 517
Months | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Rituximab-Lenalidomide vs Investigator Choice; Test type: Superiority; Hazard Ratio (HR) = 1.040, 95% CI 2-sided [0.775 to 1.395]

6. Secondary Outcome: Time to Next Anti-Lymphoma Treatment (TTNLT)
Description: Time to Next Lymphoma Treatment (TTNLT) was measured from the date of randomization to the date of the first documented administration of any new anti-lymphoma treatment (such as chemotherapy, radiotherapy, radio-immunotherapy, or immunotherapy). Participants who continued to respond to treatment or who were lost to follow-up were considered censored on their last visit date. Participants who died (due to any cause) before receiving a new anti-lymphoma treatment were included in the statistical analysis, with death being counted as an event. Based on Kaplan-Meier estimates.
Time Frame: From the date of randomization to the date of the first documented administration of any new anti-lymphoma treatment (up to approximately 140 months).
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab-Lenalidomide | Investigator Choice
Number analyzed (Participants) | 513 | 517
Months | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Rituximab-Lenalidomide vs Investigator Choice; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.809, 95% CI 2-sided [0.651 to 1.006]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from randomization to study completion (up to approximately 144 months). SAEs and Other AEs were assessed from first dose to 28 days post the last dose (up to approximately an average of 25 months and a maximum of 33 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication. The data for the Investigator Choice chemotherapy arms, previously grouped together, presented separately for each specific chemotherapy treatment that participants received.
Groups:
- Investigator Choice Rituximab-CHOP: Six cycles of R-CHOP in 21 day cycles followed by two 21 day cycles of 375 mg/m^2 rituximab and 7 weeks later responding patients continue with 375 mg/m^2 rituximab every 8 weeks for 12 cycles.
- Investigator Choice Rituximab-CVP: Eight cycles of R-CVP in 21 day cycles; and 7 weeks later responding patients continue with 375 mg/m^2 rituximab every 8 weeks for 12 cycles.
- Investigator Choice Rituximab-Bendamustine: Rituximab 375 mg/m^2 (day 1) plus bendamustine 90 mg/m^2 (days 1 + 2) every 28 days for six cycles; and 8 weeks later responding patients continue with 375 mg/m^2 rituximab every 8 weeks for 12 cycles.
Arm/Group | Rituximab-Lenalidomide | Investigator Choice Rituximab-CHOP | Investigator Choice Rituximab-CVP | Investigator Choice Rituximab-Bendamustine
All-Cause Mortality (participants affected / at risk) | 88/513 | 71/372 | 7/28 | 12/117
Serious Adverse Events (participants affected / at risk) | 181/507 | 109/365 | 7/26 | 32/112
Other Adverse Events (participants affected / at risk) | 496/507 | 351/365 | 26/26 | 108/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab-Lenalidomide (N=507) | Investigator Choice Rituximab-CHOP (N=365) | Investigator Choice Rituximab-CVP (N=26) | Investigator Choice Rituximab-Bendamustine (N=112)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 9 | 17 | 1 | 6
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 3 | 0 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0 | 1
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 2 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 1 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1 | 0 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0 | 0 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 1 | 0
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIORENAL SYNDROME (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIOTOXICITY (Cardiac disorders) | 0 | 1 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 1 | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0 | 0
SINUS NODE DYSFUNCTION (Cardiac disorders) | 0 | 1 | 0 | 0
BRUGADA SYNDROME (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
GASTROINTESTINAL MALFORMATION (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
HYPERTHYROIDISM (Endocrine disorders) | 0 | 1 | 0 | 0
CATARACT (Eye disorders) | 1 | 0 | 0 | 0
PAPILLOEDEMA (Eye disorders) | 1 | 0 | 0 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 3 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1 | 0 | 0
ASCITES (Gastrointestinal disorders) | 1 | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 2 | 0 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 3 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 4 | 3 | 0 | 0
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
FAECALOMA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 0 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0
HERNIAL EVENTRATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 2 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 3 | 0 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
POOR DENTAL CONDITION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 1
SUBILEUS (Gastrointestinal disorders) | 1 | 2 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 2 | 0 | 1
ADVERSE DRUG REACTION (General disorders) | 1 | 0 | 0 | 0
ASTHENIA (General disorders) | 2 | 0 | 0 | 0
CARDIAC DEATH (General disorders) | 0 | 1 | 0 | 0
CHEST PAIN (General disorders) | 2 | 2 | 1 | 0
FACE OEDEMA (General disorders) | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 0 | 0 | 1
FOREIGN BODY REACTION (General disorders) | 0 | 1 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 | 0 | 0 | 0
HYPERTHERMIA (General disorders) | 1 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0 | 0
MALAISE (General disorders) | 1 | 1 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 1 | 0
PYREXIA (General disorders) | 13 | 2 | 0 | 1
STRANGULATED HERNIA (General disorders) | 0 | 1 | 0 | 0
BILIARY DILATATION (Hepatobiliary disorders) | 1 | 0 | 0 | 0
BILIARY OBSTRUCTION (Hepatobiliary disorders) | 0 | 1 | 0 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 2 | 0 | 0 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0 | 0 | 0
ANAPHYLACTIC SHOCK (Immune system disorders) | 2 | 0 | 0 | 0
ANAPHYLACTOID REACTION (Immune system disorders) | 1 | 0 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 1 | 1 | 0 | 0
APPENDICITIS (Infections and infestations) | 2 | 0 | 0 | 0
BACTERIAL SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0
BACTERIURIA (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHIOLITIS (Infections and infestations) | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 2 | 1 | 0 | 0
CAMPYLOBACTER SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 1 | 0 | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
DEVICE RELATED SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
ENTEROBACTER SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
FUSOBACTERIUM INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
GANGRENE (Infections and infestations) | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 1
GENITAL HERPES SIMPLEX (Infections and infestations) | 0 | 1 | 0 | 0
H1N1 INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0
HEPATITIS E (Infections and infestations) | 1 | 0 | 0 | 0
HERPES OPHTHALMIC (Infections and infestations) | 0 | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 1 | 0 | 0
HUMAN EHRLICHIOSIS (Infections and infestations) | 0 | 0 | 0 | 1
INFECTION (Infections and infestations) | 1 | 2 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 2 | 1 | 0
LARGE INTESTINE INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
MENINGITIS (Infections and infestations) | 0 | 0 | 0 | 1
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0 | 0
PARONYCHIA (Infections and infestations) | 1 | 0 | 0 | 0
PERITONITIS (Infections and infestations) | 2 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0
PILONIDAL DISEASE (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 | 2 | 0 | 0
PNEUMONIA (Infections and infestations) | 11 | 6 | 0 | 3
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 2 | 0 | 0 | 0
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA VIRAL (Infections and infestations) | 1 | 0 | 0 | 0
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0
PSEUDOMONAS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 1 | 0 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 2 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 2 | 1 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 2 | 2 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
TONSILLITIS (Infections and infestations) | 1 | 0 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 5 | 1 | 0 | 0
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1 | 0 | 0 | 0
UROSEPSIS (Infections and infestations) | 1 | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
WOUND INFECTION BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 0 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
AORTIC INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
CHEST INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 9 | 1 | 0 | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 0 | 0 | 0 | 1
FIBRIN D DIMER INCREASED (Investigations) | 1 | 0 | 0 | 0
TROPONIN INCREASED (Investigations) | 1 | 0 | 0 | 0
TROPONIN T INCREASED (Investigations) | 1 | 0 | 0 | 0
URINE OUTPUT DECREASED (Investigations) | 0 | 0 | 0 | 1
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
CHONDROCALCINOSIS (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 0 | 4
BENIGN NEOPLASM OF EPIDIDYMIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BENIGN RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
CLEAR CELL RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
COLORECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
GALLBLADDER ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 1 | 6
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA OF THE TONGUE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 0 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 2 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 1 | 0 | 0
MIGRAINE WITH AURA (Nervous system disorders) | 0 | 1 | 0 | 0
OPTIC NEURITIS (Nervous system disorders) | 2 | 0 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 1 | 0 | 0
SEIZURE (Nervous system disorders) | 1 | 0 | 0 | 0
SPEECH DISORDER (Nervous system disorders) | 1 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 | 0 | 1 | 0
DEVICE BREAKAGE (Product Issues) | 1 | 0 | 0 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0
CONVERSION DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 0
MANIA (Psychiatric disorders) | 0 | 0 | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 | 2 | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1 | 0 | 0
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 | 1 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 5 | 1 | 0 | 0
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0 | 0
CYSTOCELE (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
PENILE ADHESION (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 0 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
CAPILLARITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
CUTANEOUS VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
HYPERSENSITIVITY VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 10 | 0 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
VASCULAR PURPURA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
UMBILICAL HERNIA REPAIR (Surgical and medical procedures) | 0 | 1 | 0 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 | 0 | 0 | 0
AORTIC DISSECTION (Vascular disorders) | 2 | 0 | 0 | 0
ARTERIAL THROMBOSIS (Vascular disorders) | 1 | 0 | 0 | 0
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 | 0 | 0 | 0
ARTERITIS (Vascular disorders) | 1 | 0 | 0 | 0
BLEEDING VARICOSE VEIN (Vascular disorders) | 0 | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 1 | 0 | 1
HAEMATOMA (Vascular disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0
PHLEBITIS (Vascular disorders) | 1 | 2 | 0 | 0
PHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0 | 0
SUPERFICIAL VEIN THROMBOSIS (Vascular disorders) | 2 | 0 | 0 | 0
THROMBOSIS (Vascular disorders) | 1 | 0 | 0 | 0
VASCULITIS (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab-Lenalidomide (N=507) | Investigator Choice Rituximab-CHOP (N=365) | Investigator Choice Rituximab-CVP (N=26) | Investigator Choice Rituximab-Bendamustine (N=112)
ANAEMIA (Blood and lymphatic system disorders) | 25 | 44 | 3 | 8
LEUKOPENIA (Blood and lymphatic system disorders) | 22 | 47 | 2 | 7
LYMPHOPENIA (Blood and lymphatic system disorders) | 7 | 19 | 1 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 199 | 172 | 7 | 25
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 17 | 14 | 0 | 11
PALPITATIONS (Cardiac disorders) | 7 | 9 | 0 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 77 | 29 | 2 | 12
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 37 | 45 | 1 | 6
CONSTIPATION (Gastrointestinal disorders) | 179 | 109 | 13 | 43
DIARRHOEA (Gastrointestinal disorders) | 184 | 50 | 6 | 37
DYSPEPSIA (Gastrointestinal disorders) | 26 | 19 | 2 | 7
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 18 | 15 | 0 | 7
NAUSEA (Gastrointestinal disorders) | 100 | 128 | 7 | 72
STOMATITIS (Gastrointestinal disorders) | 15 | 26 | 1 | 9
VOMITING (Gastrointestinal disorders) | 32 | 61 | 2 | 31
ASTHENIA (General disorders) | 144 | 129 | 6 | 5
CHILLS (General disorders) | 20 | 2 | 1 | 11
FATIGUE (General disorders) | 116 | 67 | 6 | 73
INFLUENZA LIKE ILLNESS (General disorders) | 18 | 5 | 0 | 7
MALAISE (General disorders) | 11 | 8 | 0 | 6
MUCOSAL INFLAMMATION (General disorders) | 15 | 19 | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 68 | 31 | 4 | 12
PAIN (General disorders) | 9 | 9 | 2 | 4
PYREXIA (General disorders) | 90 | 43 | 4 | 23
BRONCHITIS (Infections and infestations) | 83 | 79 | 5 | 6
CONJUNCTIVITIS (Infections and infestations) | 15 | 23 | 2 | 4
FUNGAL INFECTION (Infections and infestations) | 5 | 3 | 2 | 3
GASTROENTERITIS (Infections and infestations) | 24 | 10 | 2 | 1
HERPES ZOSTER (Infections and infestations) | 8 | 14 | 0 | 11
INFLUENZA (Infections and infestations) | 23 | 17 | 2 | 2
NASOPHARYNGITIS (Infections and infestations) | 87 | 42 | 2 | 8
PHARYNGITIS (Infections and infestations) | 19 | 17 | 2 | 2
RHINITIS (Infections and infestations) | 56 | 34 | 0 | 0
SINUSITIS (Infections and infestations) | 42 | 20 | 2 | 11
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 48 | 22 | 5 | 28
URINARY TRACT INFECTION (Infections and infestations) | 44 | 27 | 0 | 9
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 58 | 25 | 1 | 29
LYMPHOCYTE COUNT DECREASED (Investigations) | 4 | 6 | 2 | 2
WEIGHT DECREASED (Investigations) | 19 | 13 | 2 | 9
WEIGHT INCREASED (Investigations) | 8 | 7 | 2 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 14 | 44 | 0 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 19 | 14 | 1 | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 79 | 52 | 4 | 24
BACK PAIN (Musculoskeletal and connective tissue disorders) | 75 | 49 | 5 | 11
BONE PAIN (Musculoskeletal and connective tissue disorders) | 22 | 37 | 1 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 70 | 16 | 2 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 73 | 16 | 2 | 12
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 39 | 15 | 2 | 6
DIZZINESS (Nervous system disorders) | 45 | 17 | 0 | 20
DYSGEUSIA (Nervous system disorders) | 23 | 24 | 0 | 5
HEADACHE (Nervous system disorders) | 66 | 31 | 3 | 25
HYPOAESTHESIA (Nervous system disorders) | 8 | 8 | 0 | 6
NEUROPATHY PERIPHERAL (Nervous system disorders) | 35 | 72 | 2 | 6
PARAESTHESIA (Nervous system disorders) | 37 | 46 | 3 | 8
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 18 | 21 | 3 | 5
ANXIETY (Psychiatric disorders) | 27 | 24 | 0 | 11
DEPRESSION (Psychiatric disorders) | 20 | 21 | 2 | 8
INSOMNIA (Psychiatric disorders) | 31 | 34 | 3 | 21
COUGH (Respiratory, thoracic and mediastinal disorders) | 104 | 44 | 4 | 20
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 55 | 33 | 5 | 13
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 25 | 14 | 1 | 10
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 2 | 3
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 0 | 8
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 | 39 | 2 | 4
DRY SKIN (Skin and subcutaneous tissue disorders) | 44 | 13 | 0 | 4
ERYTHEMA (Skin and subcutaneous tissue disorders) | 38 | 9 | 2 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 18 | 4 | 2 | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 86 | 22 | 3 | 10
RASH (Skin and subcutaneous tissue disorders) | 141 | 22 | 1 | 19
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 19 | 5 | 1 | 6
HOT FLUSH (Vascular disorders) | 16 | 5 | 0 | 6
HYPERTENSION (Vascular disorders) | 23 | 13 | 2 | 9
HYPOTENSION (Vascular disorders) | 16 | 5 | 2 | 1
PHLEBITIS (Vascular disorders) | 2 | 4 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT01476787/Prot_SAP_000.pdf